CLINICAL TRIAL: NCT02378974
Title: A Randomized, Double-blind, Placebo-controlled, Phase I/IIa Clinical Trial for Evaluation of Safety and Potential Therapeutic Effects After Intravenous Transplantation of Human Umbilical Cord-derived Mesenchymal Stem Cells in Patients With Cerebral Infarction Disease
Brief Title: Evaluation of the Safety and Potential Therapeutic Effects of Cordstem-ST in Patients With Cerebral Infarction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHABiotech CO., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHA-CST-101
Record Dates: First submitted 2015-02-16; First posted 2015-03-04 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2019-11

CONDITIONS: Cerebral Infarction
Keywords: Cerebral Infarction; Mesenchymal Stem Cells; Stroke
MeSH Terms: conditions — Cerebral Infarction; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Other): Cordstem-ST cells or Placebo on day 0
  Interventions: Biological: Cordstem-ST; Biological: Placebo
- Cohort 2 (Other): Cordstem-ST cells or Placebo on day 0 and day 7
  Interventions: Biological: Cordstem-ST; Biological: Placebo

INTERVENTIONS:
Biological: Cordstem-ST
Biological: Placebo

SUMMARY:
The objective of the study is to evaluate the safety and the potential therapeutic effects per dose of Cordstem-ST Intravenous Transplantation in Cerebral Infarction subjects

DETAILED DESCRIPTION:
Cohort 1 : Cordstem-ST cells or Placebo on day 0 Cohort 2: Cordstem-ST cells or Placebo on day 0 and day 7

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects between 19 to 80 years of age (inclusive) at the time of screening visit
2. Subjects who are able to receive intravenous Cordstem-ST Transplantation within 7 days (168 hours) of stroke onset
3. Subjects with diagnosis of Cerebral Infarction confirmed by the following criteria assessed at the screening visit

   * NIHSS score between 5 and 20 (inclusive)
   * Acute ischemic lesion involving anterior circulation territory identified in the diffusion weighted MRI
4. Signed informed consent

Exclusion Criteria

1. History of intracranial hemorrhage
2. Subjects who are suspected to undergo endarterectomy during the study period. Subjects who received the former procedures not due to cerebral infarction more than 3 months ago, are eligible.
3. Subjects with hemorrhagic transformation on brain images, except for petechial hemorrhage ('H1' according to the ECASS classification)
4. Subjects at the high risk of developing brain herniation
5. History of dementia
6. History of epilepsy
7. Subjects who have been treated or diagnosed with schizophrenia, depression, or bipolar disorder within the past 6 months
8. Subjects with recent (≤3 months) myocardial infarction or stroke other than the index stroke.
9. Subjects must not have the following conditions in laboratory tests

   * ALT or AST: More than 2.5 times the upper limit of normal
   * Serum creatinine: More than 1.5 times the upper limit of normal
   * Total bilirubin: More than 2.5 times the upper limit of normal
   * Platelet count: less than lower limit of narmal
10. Subjects who are HBV, HCV, HIV, VDRL positive
11. Subjects in poor general condition due to medical conditions or subjects with severe cardiovascular, gastrointestinal, pulmonary, endocrinologic diseases
12. Subjects with active lung diseases, based on chest X-ray
13. Subjects with abnormal coagulopathic conditions (thrombocytopenia, congenital coagulopathy, etc.). Medical use of oral anticoagulants is permitted.
14. Subjects with known allergies to protein products (Bovine serum) used in the cell production process.
15. Subjects with history of pulmonary embolism or deep vein thrombosis
16. Subjects with history of malignancy
17. Pregnant or lactating women
18. Women of childbearing age who reject to practice contraception with one of the following methods

    * Use a condom
    * Use of contraceptive (oral, dermal, or injectable)
    * Use an intra-uterine contraceptive device
19. Subjects with a history of alcohol abuse (>30g/day) or drug abuse
20. Subjects who cannot undergo MRI scanning
21. Subjects who cannot conduct the scheduled monitoring visits
22. Subjects who is determined to be inappropriate by the investigators

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of TEAEs | 6 month
  Number of treatment related-adverse events during the study period

SECONDARY OUTCOMES:
Improvement in clinical function as assessed by mRS | 6 month
  Modified Rankin Score (mRS) compared to baseline at 6 months
Improvement in clinical function as assessed by NIHSS | 6 month
  National Institute of Health Stroke Scale (NIHSS) compared to baseline at 6 months
Improvement in clinical function as assessed by BI | 6 month
  Barthel Index (BI) compared to baseline at 6 months
Improvement in clinical function as assessed by Brain MRI tratogram | 6 month
  Brain MRI tratogram compared to baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ok Joon Kim, Principal Investigator — CHA University Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea